CLINICAL TRIAL: NCT01839994
Title: Phase III Clinical Trial on Conventionally Fractionated Conformal Radiotherapy (CF-CRT) Versus CF-CRT Combined With High-dose-rate Brachytherapy or Stereotactic Body Radiotherapy for Intermediate and High-risk Prostate Cancer.
Brief Title: Conformal Radiotherapy (CRT) Alone Versus CRT Combined With HDR BT or Stereotactic Body Radiotherapy for Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRT/BT/SBRT-COI-02
Record Dates: First submitted 2013-04-22; First posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer,; high-dose-rate brachytherapy boost,; stereotactic body radiotherapy boost,; conformal radiotherapy,; randomized trial
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CF-CRT combined with BT or SBRT boost (Experimental): Conventionally fractionated CRT (IMRT or Rapid Arc) to the TD of 50 Gy, 2.0 Gy d fx, 5 days a week over the period of 5 weeks AND two 10 Gy fractions of real- time HDR brachytherapy OR CRT combined with two stereotactic body radiotherapy boosts of 10 Gy per fraction delivered with dynamic SBRT technique (IMRT or Rapid Arc).
  The choice between two ways of delivering radiation dose to the boost volume will be based solely on clinical criteria, decision made by interdisciplinary team, according to the institutional protocol (in non-randomized fashion).
  Hormonal treatment: three months of neoadjuvant androgen deprivation (MAB -maximal androgen blockade) in all patients. Long-term (3 years) of adjuvant hormonotherapy (LHRH agonists only) in high risk patients.
  Interventions: Radiation: CF-CRT combined with BT or SBRT boost.; Drug: Hormonal treatment (neoadjuvant androgen deprivation)
- CF-CRT alone (Active Comparator): Conventionally fractionated external beam conformal radiotherapy (IMRT or Rapid Arc) to the prostate and seminal vesicles (intermediate risk group) or to the prostate, SV and pelvic lymph nodes (high risk group) to the total dose of 50 Gy in 2.0 Gy per fraction, 5 days a week over the period of 5 weeks, followed by a boost to the prostate (26 or 28 Gy in 2.0 Gy per fraction 5 days a week over the period of 2.5 weeks) to the total dose of 76 or 78 Gy (intermediate or high risk group of patients, respectively).
  Hormonal treatment: three months of neoadjuvant androgen deprivation (MAB -maximal androgen blockade) in all patients. Long-term (3 years) of adjuvant hormonotherapy (LHRH agonists only) in high risk patients.
  Interventions: Radiation: CF-CRT alone; Drug: Hormonal treatment (neoadjuvant androgen deprivation)

INTERVENTIONS:
Radiation: CF-CRT combined with BT or SBRT boost. — CF-CRT to the prostate and SV (IM risk group) or to the prostate, SV and LN (high risk group) to the TD of 50 Gy, 2.0 Gy d fx, 5 days a week over the period of 5 weeks AND A. Two 10 Gy fractions of HDR BT 1-7 d. before external beam radiotherapy and one 1-7 d. after external beam radiotherapy OR B. Two stereotactic body radiotherapy (SBRT) fractions of 10 Gy to the prostate (CTV boost) delivered with dynamic SBRT technique (IMRT or Rapid Arc). First and second fraction of SBRT boost is scheduled 1-7 d. before and 1-7 d. after the start of conventionally fractionated radiotherapy, respectively.
  Arms: CF-CRT combined with BT or SBRT boost
Radiation: CF-CRT alone — Conventionally fractionated EB-CRT (IMRT or Rapid Arc) to the TD of 50 Gy, followed by a boost to the prostate (26 or 28 Gy in 2.0 Gy per fraction 5 days a week over the period of 2.5 weeks) to the total dose of 76 or 78 Gy (intermediate or high risk group of patients, respectively).of 50 Gy in 2.0 Gy per fraction, 5 days a week over the period of 5 weeks, followed by a boost to the prostate (26 or 28 Gy in 2.0 Gy per fraction 5 days a week over the period of 2.5 weeks) to the total dose of 76 or 78 Gy (intermediate or high risk group of patients, respectively).
  Arms: CF-CRT alone
Drug: Hormonal treatment (neoadjuvant androgen deprivation) — Hormonal treatment: three months of neoadjuvant androgen deprivation (MAB -maximal androgen blockade) in all patients. Long-term (3 years) of adjuvant hormonotherapy (LHRH agonists only) in high risk patients.

SUMMARY:
The purpose of this study is to compare the outcomes of conventionally fractionated conformal radiotherapy with CF-CRT combined with either high-dose-rate brachytherapy or stereotactic body radiotherapy for intermediate or high-risk prostate cancer patients.

DETAILED DESCRIPTION:
Prostate cancer is considered as a disease with relatively slow natural course and good clinical prognosis. Such description, however, does not well refer to intermediate and high-risk cases where long-term rate of biochemical progression remains not satisfactory, and the available treatment modalities entail a considerable morbidity. Over the last decade several competitive therapeutic approaches have evolved in curative treatment for intermediate and high-risk prostate cancer. The use of intensity-modulated radiation therapy (IMRT) made possible to escalate the total dose to the prostate without excessive toxicity.

Based on assumption of low value of low α/β value for adenocarcinoma of prostate, there is a potential of escalating the biological dose to the tumor with higher dose per fraction. High-dose-rate brachytherapy (HDR-BT) is one of the options, with the ability to conform radiation dose to the prostate with sharp dose gradient adjacent to critical organs. An increasing number of studies suggest its usefulness as a boost in intermediate and high risk disease. The randomized trial conducted in UK compared external beam radiotherapy (EBRT) alone with EBRT and HDR brachytherapy as a boost. Combining EBRT with HDR BT - boost resulted in significantly higher relapse-free-survival (RFS) with comparable incidence of severe late toxicity. However, the total dose used in EBRT alone - arm and radiotherapy technique may be considered suboptimal according to current standards.

Stereotactic body radiotherapy (SBRT) may be an interesting alternative to HDR brachytherapy, not requiring implantation of multiple catheters and anesthesia. SBRT boost for advanced localized prostate cancer has the potential to reduce toxicity while escalating the dose. First results of trials combining conventional irradiation with hypofractionated stereotactic boost and institutional pilot results gave promising outcome.

The comparison of these modalities of radiation therapy for prostate cancer will be performed in the current phase III trial study.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven adenocarcinoma of the prostate
2. Clinical stage T1-T3a (Intermediate or high risk features according to NCCN criteria)
3. No evidence of nodal or distant spread as determined by chest X-ray, bone scan and abdominal ultrasound or CT-scan or other investigations such as Positron Emission Tomography [PET] scan if required
4. No evidence of bulky spread beyond the capsule of the prostate, no seminal vesicle involvement assessed by TRUS or MRI of pelvis.
5. Good performance status (ZUBROD <2, Karnofsky index >=80%).
6. No contradictions for spinal anesthesia.
7. No contradictions for hormonal treatment (androgen deprivation).
8. Adequate bone marrow, renal and liver function.
9. Life expectancy in excess of 5 years.
10. No prior malignancy, except basal or squamous cell skin cancer.
11. Informed consent for participation in the study (confirmed by the signature together with the standard medical consent form for radiotherapy within the pelvis)

Exclusion Criteria:

1. Different histology than adenocarcinoma.
2. Previous or concurrent malignancy, with the exception of basal cell carcinoma of the skin.
3. Locally advanced disease: bulky T3a and/or T3b.
4. Presence of metastatic disease (nodal and/or distant).
5. PSA >100ng/ml
6. Any previous therapy other than hormonal treatment.
7. Concurrent uncontrolled medical conditions.
8. Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
9. Withdrawal of informed consent.

   -

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from biochemical failure (FFBF) | 3 years
  according to Phoenix definition (rise of PSA level of 2 ng/ml over the absolute nadir)

SECONDARY OUTCOMES:
Freedom from local relapse | 3 years
Freedom from loco-regional relapse | 3 years
Freedom from distant metastases | 3 years
Time of occurrence, incidence and severity of acute normal tissue reactions as measured according to CTCAE v4.0 and RTOG/EORTC scoring system | 3 months
Time of occurrence, incidence and severity late normal tissue reactions as measured according to CTCAE v4.0 and RTOG/EORTC scoring system | 3 years
Overall survival | 5 years
Progression-free survival | 3 years

OTHER OUTCOMES:
Identification of molecular and biochemical predictors of response to external beam radiotherapy and brachytherapy or SBRT boost as compared to external beam radiotherapy alone | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rafał Suwiński, MD, PhD, Principal Investigator — Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Poland
Locations (1):
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Gliwice Branch, Gliwice, Silesian Voivodeship, Poland

REFERENCES:
- [Background] Zelefsky MJ, Chan H, Hunt M, Yamada Y, Shippy AM, Amols H. Long-term outcome of high dose intensity modulated radiation therapy for patients with clinically localized prostate cancer. J Urol. 2006 Oct;176(4 Pt 1):1415-9. doi: 10.1016/j.juro.2006.06.002. PMID 16952647
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Pieters BR, de Back DZ, Koning CC, Zwinderman AH. Comparison of three radiotherapy modalities on biochemical control and overall survival for the treatment of prostate cancer: a systematic review. Radiother Oncol. 2009 Nov;93(2):168-73. doi: 10.1016/j.radonc.2009.08.033. Epub 2009 Sep 11. PMID 19748692
- [Background] Martinez AA, Gustafson G, Gonzalez J, Armour E, Mitchell C, Edmundson G, Spencer W, Stromberg J, Huang R, Vicini F. Dose escalation using conformal high-dose-rate brachytherapy improves outcome in unfavorable prostate cancer. Int J Radiat Oncol Biol Phys. 2002 Jun 1;53(2):316-27. doi: 10.1016/s0360-3016(02)02733-5. PMID 12023135
- [Background] Martinez AA, Gonzalez J, Ye H, Ghilezan M, Shetty S, Kernen K, Gustafson G, Krauss D, Vicini F, Kestin L. Dose escalation improves cancer-related events at 10 years for intermediate- and high-risk prostate cancer patients treated with hypofractionated high-dose-rate boost and external beam radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):363-70. doi: 10.1016/j.ijrobp.2009.10.035. PMID 21195875
- [Background] Hoskin PJ, Rojas AM, Bownes PJ, Lowe GJ, Ostler PJ, Bryant L. Randomised trial of external beam radiotherapy alone or combined with high-dose-rate brachytherapy boost for localised prostate cancer. Radiother Oncol. 2012 May;103(2):217-22. doi: 10.1016/j.radonc.2012.01.007. Epub 2012 Feb 16. PMID 22341794
- [Background] Miralbell R, Molla M, Rouzaud M, Hidalgo A, Toscas JI, Lozano J, Sanz S, Ares C, Jorcano S, Linero D, Escude L. Hypofractionated boost to the dominant tumor region with intensity modulated stereotactic radiotherapy for prostate cancer: a sequential dose escalation pilot study. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):50-7. doi: 10.1016/j.ijrobp.2009.07.1689. Epub 2009 Nov 10. PMID 19910135
- [Background] Quon H, Cheung PC, Loblaw DA, Morton G, Pang G, Szumacher E, Danjoux C, Choo R, Kiss A, Mamedov A, Deabreu A. Quality of life after hypofractionated concomitant intensity-modulated radiotherapy boost for high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2012 Jun 1;83(2):617-23. doi: 10.1016/j.ijrobp.2011.07.005. Epub 2011 Nov 11. PMID 22079736
- [Background] Jabbari S, Weinberg VK, Kaprealian T, Hsu IC, Ma L, Chuang C, Descovich M, Shiao S, Shinohara K, Roach M 3rd, Gottschalk AR. Stereotactic body radiotherapy as monotherapy or post-external beam radiotherapy boost for prostate cancer: technique, early toxicity, and PSA response. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):228-34. doi: 10.1016/j.ijrobp.2010.10.026. Epub 2010 Dec 22. PMID 21183287
- [Background] Oermann EK, Slack RS, Hanscom HN, Lei S, Suy S, Park HU, Kim JS, Sherer BA, Collins BT, Satinsky AN, Harter KW, Batipps GP, Constantinople NL, Dejter SW, Maxted WC, Regan JB, Pahira JJ, McGeagh KG, Jha RC, Dawson NA, Dritschilo A, Lynch JH, Collins SP. A pilot study of intensity modulated radiation therapy with hypofractionated stereotactic body radiation therapy (SBRT) boost in the treatment of intermediate- to high-risk prostate cancer. Technol Cancer Res Treat. 2010 Oct;9(5):453-62. doi: 10.1177/153303461000900503. PMID 20815416